CLINICAL TRIAL: NCT00784797
Title: Comparison Between Misopristol and Pitocin After Mifepristone Preparation for Second Trimeter Abortion
Brief Title: Misopristol Versus Pitocin for Second Trimester Abortion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Assaf Ben Meir, MD, Hadassah Medical Organization
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PitocinPGMyf-HMO-CTIL
Record Dates: First submitted 2008-11-02; First posted 2008-11-04 (Estimated); Last update posted 2013-11-21 (Estimated); Status verified 2013-11

CONDITIONS: Abortion, Missed
MeSH Terms: conditions — Abortion, Missed | interventions — Mifepristone; Oxytocin

ARMS (2):
- pitocin (Active Comparator): high dose pitocin drip 48 hours after mifepristone preparation.
  Interventions: Drug: mifepristone and oxytocin
- misopristol (Active Comparator): vaginal and oral misopristol 48 hours after mifepristone preparation.
  Interventions: Drug: mifepristone and misopristol

INTERVENTIONS:
Drug: mifepristone and misopristol — 200 mg mifepristone and after 48 hours vaginal misopristol 800 mgr followed by oral misopristol 400 mgr every 3 hours for maxamum 5 doses
  Arms: misopristol
Drug: mifepristone and oxytocin — 200 mg mifepristone followed 48 hours with high dose oxytocin drip (9 unit per hour)
  Arms: pitocin

SUMMARY:
Second trimester abortion can be done surgically or medically. Medical abortion with mifepristone and misopristol is one of the common protocol, but misopristol have high rate side effect. The investigators recent study proved the efficacy of pitocin after mifepristone in second trimester abortion with minimal side effects.

Working hypothesis and aims: To compare misopristol and pitocin after mifepristone preparation in second trimester in seccess rate, interval to abortion, side effects and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* midtrimester late abortion
* midtrimester induced abortion

Exclusion Criteria:

* placenta previa
* infected abortion
* rupture of membranes
* s/p cesarean section *2 or more

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 145 (Actual)
Dates: Start 2009-01; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Success rate of abortion | 24 hours
Interval to abortion | 24 hours

SECONDARY OUTCOMES:
Side effects | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Assaf Ben-Meir, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

REFERENCES:
- [Derived] Ghosh J, Papadopoulou A, Devall AJ, Jeffery HC, Beeson LE, Do V, Price MJ, Tobias A, Tuncalp O, Lavelanet A, Gulmezoglu AM, Coomarasamy A, Gallos ID. Methods for managing miscarriage: a network meta-analysis. Cochrane Database Syst Rev. 2021 Jun 1;6(6):CD012602. doi: 10.1002/14651858.CD012602.pub2. PMID 34061352
- [Derived] Freeman MD, Porat N, Rojansky N, Elami-Suzin M, Winograd O, Ben-Meir A. Physical symptoms and emotional responses among women undergoing induced abortion protocols during the second trimester. Int J Gynaecol Obstet. 2016 Nov;135(2):154-157. doi: 10.1016/j.ijgo.2016.05.008. Epub 2016 Aug 15. PMID 27539053
- [Derived] Elami-Suzin M, Freeman MD, Porat N, Rojansky N, Laufer N, Ben-Meir A. Mifepristone followed by misoprostol or oxytocin for second-trimester abortion: a randomized controlled trial. Obstet Gynecol. 2013 Oct;122(4):815-820. doi: 10.1097/AOG.0b013e3182a2dcb7. PMID 24084539